CLINICAL TRIAL: NCT04598724
Title: Addressing Barriers to Palliative Care Use in Bladder Cancer Through Better Understanding of Knowledge and Belief Development
Brief Title: Addressing Barriers to Palliative Care Use in Bladder Cancer
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-20809
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Muscle-Invasive Bladder Carcinoma; Bladder Cancer Stage II; Bladder Cancer Stage III; Bladder Cancer Stage IV
Keywords: Bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bladder Cancer Patient Participants: Participants will be scheduled for one-on-one interviews that will occur over Zoom or telephone.
  Interventions: Other: Surveys
- Care Givers for Bladder Cancer Patient Participants: Participants will be scheduled for one-on-one interviews that will occur over Zoom or telephone.
  Interventions: Other: Surveys

INTERVENTIONS:
Other: Surveys — Survey will be administered involving questions regarding knowledge and perception of palliative care.

SUMMARY:
Investigators plan to establish an in-depth understanding of knowledge and beliefs about palliative care in advanced Bladder Cancer patients and their caregivers, and to identify factors associated with positive and negative experiences with palliative care services among those who have received them.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for both patient and caregiver participants will include:
* age ≥18 years
* able to speak and read English
* cognitively able to participate in study tasks
* willing to participate in surveys, semi-structured interviews, and/or focus groups
* able to participate in either a Zoom meeting or phone interview
* able to complete an emailed or paper survey
* Patient Participants: a diagnosis of muscle-invasive or locally advanced bladder cancer (stages II-IV).

Exclusion Criteria:

* Patients and caregivers will be excluded if unable to provide verbal or written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Bladder Cancer patient participants and care givers will be recruited from the Moffitt Cancer Genitourinary Oncology clinic and the Supportive Care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Development of palliative care knowledge and beliefs | 12 Months
  Thematic analysis of interviews transcriptions to identify the themes that underpin the development of palliative care beliefs among patients with muscle invasive bladder cancer.
Proportion with accurate palliative care knowledge and beliefs | 12 Months
  Proportion of patients correctly answering each palliative care knowledge question.

SECONDARY OUTCOMES:
Association between Bladder Cancer stage and palliative care knowledge | 12 Months
  Analysis of variance calculated for the mean number of subjects with each cancer stage correctly answering each palliative care knowledge question

CONTACTS AND LOCATIONS:
Overall Officials: Scott Gilbert, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trial Search — https://moffitt.org/clinical-trials-research/clinical-trials/